CLINICAL TRIAL: NCT01899222
Title: Assessment of Prototype Hand-Held Fundus Camera
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, David Kleinman, Medical Doctor and Department Faculty, University of Rochester
Other Study IDs: HHFC 02
Record Dates: First submitted 2013-07-12; First posted 2013-07-15 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Normal Subject Population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fundus imaging: retinal photograph obtained at visit
  Interventions: Device: Handheld fundus photography

INTERVENTIONS:
Device: Handheld fundus photography — diagnostic imaging with two types of retina camera
  Other Names: imaging only

SUMMARY:
Assessment of handheld fundus images in comparison to conventional fundus camera images.

DETAILED DESCRIPTION:
This study is comparing a small handheld camera with a standard fundus camera for image quality

ELIGIBILITY:
Inclusion criteria:

* Age > 18
* The ability to give informed consent and be willing to spend up to two hours in the eye clinic during the duration of the study.
* The subjects may have a normal retina and optic nerve, or subjects may have abnormalities of the posterior pole of the retina or the optic nerve.

Exclusion criteria:

* Medical or ophthalmic instability that would create a contraindication for minimally invasive ophthalmic diagnostic testing will exclude participation as a subject.
* Ophthalmic pathology felt by the principal investigator that would make retinal imaging with standard photographs difficult or not possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmology clinic
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2015-10-08 (Actual); Study Completion 2015-10-08 (Actual)

PRIMARY OUTCOMES:
Percentage of photographs that score a "3" or higher on the grading scale | 2-3 years
  Photos will be evaluated by ophthalmologists and scored as follows:
  1. Unacceptable: cannot see fundus detail
  2. Unacceptable: fundus detail visualized, but inadequate for meaningful analysis
  3. Acceptable: fundus detail visualized enough to make general comments, with modest improvement image would be of sufficient quality for widespread use
  4. Good: fundus detail visualized, meaningful analysis possible, standard photograph superior
  5. Excellent: fundus detail visualized as well as standard photograph
  6. Superior: fundus detail of higher quality than standard photograph

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States